CLINICAL TRIAL: NCT01269970
Title: Early Metabolic Response Evaluation With 18-FDG PET-CT in Esophageal Cancer Treated With Neoadjuvant Chemoradiotherapy Followed by Esophagectomy
Brief Title: Early Metabolic Response in Locally Advanced Esophageal Cancer Undergoing Induction Chemoradiotherapy
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Other Study IDs: G.0175.03; S24640 (Registry Identifier: clinical trial center UZLeuven)
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: Esophageal Carcinoma (Squamous Cell Carcinoma - Adenocarcinoma)
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- locally advanced esophageal carcinoma (cT2-3N0/+)
  Interventions: Other: 18-FDG-PET-CT

INTERVENTIONS:
Other: 18-FDG-PET-CT

SUMMARY:
Early metabolic response evaluation may predict clinical and histopathological response after neoadjuvant chemotherapy. Its value in neoadjuvant chemoradiotherapy (CRT) is unknown. Our aim was to assess the value of early metabolic response after one cycle of chemotherapy using 18-FDG-PET-CT to predict pathological response and outcome in cT2-4 N0/+ esophageal cancer treated by neoadjuvant CRT and esophagectomy.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced esophageal cancer (cT2-4 N0/+)

Exclusion Criteria:

* PET-CT not performed at UZLeuven
* Other tumor types
* Distant metastases (organ)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: locally advanced esophageal cancer (cT2-4 N0/+) of the esophagus (n=42) and GEJ (n=13)
Sampling Method: Probability Sample
Dates: Start 2004-01; Primary Completion 2008-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
early metabolic response to predict pathological response and outcome
  assess the value of early metabolic response with 18-FDG-PET-CT (i.e. a decrease of ≥ 35% of SUVmean) after a single cycle of chemotherapy followed by neoadjuvant CRT and esophagectomy as a tool to predict pathological response and outcome in patients with cT2-4N0/+ carcinoma of the esophagus and GE-junction (GEJ).

SECONDARY OUTCOMES:
to study correlations between early metabolic response, late metabolic response, histopathological response and outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- UZLeuven, Leuven, Vlaams-Brabant, Belgium